CLINICAL TRIAL: NCT06220240
Title: Does a Modified Training Program Affect Energy Deficiency and Sportive Performance?
Brief Title: Energy Deficiency and Athletic Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4203*929*
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Female Athlete Triad
Keywords: Energy Deficiency; Eccentric Exercise; Athletic Performans
MeSH Terms: conditions — Female Athlete Triad Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator administering the treatment and the investigator performing the evaluations will be different. The evaluator will not know about the interventions that the participants received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Training Group (Active Comparator): It is a training program that will be carried out under the supervision of a physiotherapist. There will be 3-minute breaks between sets. A training program will be applied to the athletes based on revising the training program they use in their routine with eccentric contractions.
  Interventions: Other: Modified Training Programme
- Routine Training Group (Active Comparator): The training program that the athlete uses in her normal routine will be implemented under the supervision of a physiotherapist.
  Interventions: Other: Routine Training Programme

INTERVENTIONS:
Other: Modified Training Programme — Eccentric muscle contractions and 3-minute rest breaks will be used.
  Arms: Modified Training Group
Other: Routine Training Programme — A routine training program will be used.
  Arms: Routine Training Group

SUMMARY:
Energy availability (EA) refers to the balance between daily energy intake and exercise energy expenditure. Athletically inadequate EA is defined as low energy availability (LEA). Energy deficits occur throughout life, from young athletes with a relative lack of energy in sports or the female athlete triad to older adults struggling with weight loss. Acute and/or chronic LEA can cause negative athletic and health outcomes in athletes.

It is known that LEA, as an energy saving mechanism, suppresses the reproductive system and causes disruption of the menstrual cycle, as well as causing many interrelated endocrine-related physiological consequences by changing other hormonal pathways. Menstrual dysfunction due to LEA causes various risks as it can disrupt the EC during training and competition. Therefore, low EA may contribute to poor sports performance due to detrimental endocrine effects.

Various parameters such as body mass and nutritional intake affect the performance of athletes, and LEA is frequently reported among athletes with intense training programs. LEA combined with high training volumes; It can cause negative consequences such as impaired protein synthesis/degradation rate, impaired hormonal and training response, increased risk of fatigue, and these can lead to decreased performance. Resting metabolic rate, which indicates the energy expended for basic body functions, is considered a potential objective indicator of energy availability.

Regulation of dietary energy intake in the management of LEA in athletes covers a wide area in the literature. However, LEA is caused not only by a deficiency in energy intake but also by an excess in energy expenditure. In the light of this information, the aim of the study is to examine the acute period effects of the training program in which exercise energy expenditure is reduced in terms of energy availability and athletic performance.

DETAILED DESCRIPTION:
Voluntary participants who have been diagnosed with energy deficiency will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into two groups. Study groups will be as follows: a) Modified Training, b) Routine Training.

ELIGIBILITY:
Inclusion Criteria:

* 18- 35 years old female gender
* Body mass index being less than 18.50-24.99 kg/m2
* Having a energy deficiency
* Been interested in basketball professionally for at least one year
* Must be training with the team at least 3 days a week
* Performance levels should be 3-4

Exclusion Criteria:

* Having a history of any fracture in the last year
* Having had a sports injury in the last 8 months
* Having had an infectious disease in the last 6 months being a smoker
* Getting 2 or more points from the SCOFF survey
* Having been using any medication regularly for the last 6 months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Woman
Enrollment: 78 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Energy Availability | change from baseline pain at 2 weeks
  The underlying etiology of Relative Energy Deficiency in Sports is low energy availability, which occurs when dietary energy intake is inadequate for an athlete's physical activity level.
  "Energy availability = Energy Intake (kcal) - Exercise Energy Expenditure (kcal/fat - free mass [fat free mass; kg])"
Relative Energy Deficiency in Sports Clinical Assessment Tool (RED-S CAT) | 3 times for 2 weeks
  It is a clinical assessment tool used to evaluate athletes or active individuals with suspected low energy availability and serves as a guide for clinicians and coaches in return-to-play decisions.
Running Performance Analysis - Biomechanics | 3 times for 2 weeks
  Performance analysis will be performed on a 10-meter platform with DigitSole in order to evaluate the biomechanics.
Running Performance Analysis - Running Speed | 3 times for 2 weeks
  Performance analysis will be performed on a 10-meter platform with DigitSole in order to evaluate the running speed.
Running Performance Analysis - Economy of the Running | 3 times for 2 weeks
  Performance analysis will be performed on a 10-meter platform with DigitSole in order to evaluate the economy of the athlete's running activity.

SECONDARY OUTCOMES:
Gonadotropin-Releasing Hormone Levels | 3 times for 2 weeks
  Low energy availability is a condition that suppresses and disrupts hormonal function.
Adrenocorticotropic Hormone Levels | 3 times for 2 weeks
  Low energy availability is a condition that suppresses and disrupts hormonal function.
thyroid stimulating Hormone Levels | 3 times for 2 weeks
  Low energy availability is a condition that suppresses and disrupts hormonal function.
Luteinizing Hormone Levels | 3 times for 2 weeks
  Low energy availability is a condition that suppresses and disrupts hormonal function.
Follicle-stimulating Hormone Levels | 3 times for 2 weeks
  Low energy availability is a condition that suppresses and disrupts hormonal function.
Vertical Jump | 3 times for 2 weeks
  The athlete will be positioned in a standing vertical position, with his feet shoulder-width apart. The athlete will reach the highest point he can in the vertec and this point will be considered the zero point. It will be asked to jump 3 times on a force plate to the highest level it can jump and the highest value will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Loucks AB, Kiens B, Wright HH. Energy availability in athletes. J Sports Sci. 2011;29 Suppl 1:S7-15. doi: 10.1080/02640414.2011.588958. Epub 2011 Jul 28. PMID 21793767
- [Background] Mountjoy M, Sundgot-Borgen JK, Burke LM, Ackerman KE, Blauwet C, Constantini N, Lebrun C, Lundy B, Melin AK, Meyer NL, Sherman RT, Tenforde AS, Klungland Torstveit M, Budgett R. IOC consensus statement on relative energy deficiency in sport (RED-S): 2018 update. Br J Sports Med. 2018 Jun;52(11):687-697. doi: 10.1136/bjsports-2018-099193. No abstract available. PMID 29773536
- [Background] De Souza MJ, Nattiv A, Joy E, Misra M, Williams NI, Mallinson RJ, Gibbs JC, Olmsted M, Goolsby M, Matheson G; Female Athlete Triad Coalition; American College of Sports Medicine; American Medical Society for Sports Medicine; American Bone Health Alliance. 2014 Female Athlete Triad Coalition consensus statement on treatment and return to play of the female athlete triad: 1st International Conference held in San Francisco, CA, May 2012, and 2nd International Conference held in Indianapolis, IN, May 2013. Clin J Sport Med. 2014 Mar;24(2):96-119. doi: 10.1097/JSM.0000000000000085. PMID 24569429
- [Background] Loucks AB, Stachenfeld NS, DiPietro L. The female athlete triad: do female athletes need to take special care to avoid low energy availability? Med Sci Sports Exerc. 2006 Oct;38(10):1694-700. doi: 10.1249/01.mss.0000239397.01203.83. No abstract available. PMID 17019289
- [Background] Heikura IA, Burke LM, Bergland D, Uusitalo ALT, Mero AA, Stellingwerff T. Impact of Energy Availability, Health, and Sex on Hemoglobin-Mass Responses Following Live-High-Train-High Altitude Training in Elite Female and Male Distance Athletes. Int J Sports Physiol Perform. 2018 Sep 1;13(8):1090-1096. doi: 10.1123/ijspp.2017-0547. Epub 2018 Sep 13. PMID 29431548
- [Background] Joy E, De Souza MJ, Nattiv A, Misra M, Williams NI, Mallinson RJ, Gibbs JC, Olmsted M, Goolsby M, Matheson G, Barrack M, Burke L, Drinkwater B, Lebrun C, Loucks AB, Mountjoy M, Nichols J, Borgen JS. 2014 female athlete triad coalition consensus statement on treatment and return to play of the female athlete triad. Curr Sports Med Rep. 2014 Jul-Aug;13(4):219-32. doi: 10.1249/JSR.0000000000000077. PMID 25014387
- [Background] Joy E, Kussman A, Nattiv A. 2016 update on eating disorders in athletes: A comprehensive narrative review with a focus on clinical assessment and management. Br J Sports Med. 2016 Feb;50(3):154-62. doi: 10.1136/bjsports-2015-095735. PMID 26782763
- [Background] Elliott-Sale KJ, Tenforde AS, Parziale AL, Holtzman B, Ackerman KE. Endocrine Effects of Relative Energy Deficiency in Sport. Int J Sport Nutr Exerc Metab. 2018 Jul 1;28(4):335-349. doi: 10.1123/ijsnem.2018-0127. Epub 2018 Jul 14. PMID 30008240
- [Background] Logue DM, Madigan SM, Melin A, Delahunt E, Heinen M, Donnell SM, Corish CA. Low Energy Availability in Athletes 2020: An Updated Narrative Review of Prevalence, Risk, Within-Day Energy Balance, Knowledge, and Impact on Sports Performance. Nutrients. 2020 Mar 20;12(3):835. doi: 10.3390/nu12030835. PMID 32245088